CLINICAL TRIAL: NCT01509235
Title: Exercise Coupled to Self Drainage in Pediatric Cystic Fibrosis Patients: an Open Label Cross Over Randomised Clinical Trial
Brief Title: Self Drainage in Pediatric Cystic Fibrosis Patients
Acronym: GYM-MUCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005.403
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; Lung function; physical exercise
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Exercise testing and self drainage session (Experimental)
  Interventions: Procedure: Chest physiotherapy
- 2. Chest physiotherapy (CP) session (Active Comparator)
  Interventions: Procedure: Chest physiotherapy

INTERVENTIONS:
Procedure: Chest physiotherapy — The whole exercise session consisted of three short period of exercise of 5 minutes each entirely done under the physiotherapists' supervision (FA).

SUMMARY:
In the current study, we designed a cross-over, open label, randomized controlled clinical trial that aim to investigate the superiority of physical exercise coupled with self drainage to a chest physiotherapy in stable cystic fibrosis children. We hypothesized that CF children undergoing physical exercise coupled to self drainage will increase the amount of expectorate secretions compared to conventional CP course, while being more satisfied and without worsening their pulmonary function status.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis diagnosis confirmed by 2 positive sudoriparous diagnostic tests
* Age : 7 to 17 years
* Capacity to expectorate
* Clinically stable
* Ability to pedal on a bike and to respect orders for physical session

Exclusion Criteria:

* Haemoptysis > 50ml
* Permanent non-invasive ventilation
* Respiration or digestive evolutive clinical abnormality
* Exacerbation

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
weight of sputum that was expectorated | 12 months
  The Physiotherapist collected all sputum excreted from the beginning of the session and during the first hour.

SECONDARY OUTCOMES:
patient's satisfaction | 12 months
  evaluation of FEV1 before and after the session, ii) sessions' quality (i.e. patients' cooperation), iii) patient's satisfaction. Patient's cooperation was quoted by the physiotherapist from 1 (patient refused to participate) to 5 (excellent participation). Patients' satisfaction was scored using a visual analogic scale (VAS) graduated from 0 (not satisfied at all) to 100 (totally satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Bellon, MD, Principal Investigator — Hospices Civils de Lyon

REFERENCES:
- [Derived] Reix P, Aubert F, Werck-Gallois MC, Toutain A, Mazzocchi C, Moreux N, Bellon G, Rabilloud M, Kassai B. Exercise with incorporated expiratory manoeuvres was as effective as breathing techniques for airway clearance in children with cystic fibrosis: a randomised crossover trial. J Physiother. 2012;58(4):241-7. doi: 10.1016/S1836-9553(12)70125-X. PMID 23177226